CLINICAL TRIAL: NCT06064968
Title: Effectiveness of Intermittent Bladder Catheterization (IBC) in Reducing Recurrence of Urethral Stricture Among Female Patients in Tertiary Care Hospital, Lahore: A Nurse Led Intervention
Brief Title: Effectiveness of Intermittent Bladder Catheterization (IBC) in Reducing Recurrence of Urethral Stricture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Farah Naz, Principal investigator, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: US RCT 001
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-05

CONDITIONS: Urethral Stricture
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Intervention Model Description: Intervention and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): In intervention group, researcher will explain the patient about the intermittent catheterization technique and give the practical demonstration for better patient understanding and make correction in patient's technique of intermittent bladder catheterization.
  Patient will be followed from the day of recruitment in the study after every 02 weeks by the researcher for 2 successive months.
  In every follow up session, assessment of the urinary complaints via AUA scoring, review of patient's technique of urethral catheterization in intervention group, and each patient's adherence to the intermittent bladder catheterization (IBC) will be noted
  Interventions: Other: Intermittent bladder catheterization
- Control group (Active Comparator): In control group already diagnosed cases of urethral stenosis who have undergone urethral dilatation will be followed fortnightly for AUA symptoms scoring for urinary complaints and urethral catheterization with nelton 14 Fr to exclude urethral stricture recurrence.
  Interventions: Other: Intermittent bladder catheterization

INTERVENTIONS:
Other: Intermittent bladder catheterization — Intermittent bladder catheterization will be taught and performed by intervention group twice daily.

SUMMARY:
The goal of this randomized controlled trial is to To assess the effectiveness of intermittent bladder catheterization (IBC) in reducing the recurrence of urethral stricture among females in tertiary care hospital, Lahore.

All the patient who have undergone urethral dilation by urologist will be divided into two groups i.e. intervention group and control group.

In control group already diagnosed cases of urethral stenosis who have undergone urethral dilatation will be followed fortnightly for AUA symptoms scoring for urinary complaints and urethral catheterization with nelton 14 Fr to exclude urethral stricture recurrence.

In intervention group, researcher will explain the patient about the intermittent catheterization technique and give the practical demonstration for better patient understanding and make correction in patient's technique of intermittent bladder catheterization.

Patient will be followed from the day of recruitment in the study after every 02 weeks by the researcher for 2 successive months.

In every follow up session, assessment of the urinary complaints via AUA scoring, review of patient's technique of urethral catheterization in intervention group, and each patient's adherence to the intermittent bladder catheterization (IBC) will be noted.

DETAILED DESCRIPTION:
Urethral stricture is a known pathology with significant health related issues ranging from mild lower urinary tract symptoms to severe urinary retention or even renal failure. Female urethral stricture (FUS) is under reported in literature. This low prevalence (4-18%) is due to lack of standard definition of the said disease, well-established diagnostic criteria and single effective treatment. Internationally, variety of literature is available on treatment of urethral stricture with urethral dilation, with or without intermittent catheterization, with wide range of disparity in recurrence rates (i.e. 43% with urethral dilation with IBC to 94% with urethral dilatation without IBC). On national level, urethral stricture disease is frequently seen in clinical practice, however, there is lack of any published data on disease management and follow up. Intermittent bladder catheterization is an acceptable mean to prevent recurrence and easy-to-perform by the patients themselves, this study is therefore, designed to assess whether intermittent bladder catheterization is effective or not in lowering the disease recurrence in patients with urethral stricture following urethral dilation. Aim of this study is to assess the effectiveness intermittent bladder catheterization (IBC) led by urology care nurse in reducing the rate of recurrence of urethral stricture in females following urethral dilation. A randomized controlled trial will be conducted and patients meeting inclusion criteria will be allocated in two groups by block randomization i.e. a control group and the intervention group. Duration of study will be 6 months after approval of synopsis. Females already diagnosed with urethral stricture disease, who have undergone urethral dilatation at least once by urologist, age between 35- 65 years, BMI <30, Abbreviated Mental Test Score (AMTS) between 7-10, and American Urological Association (AUA) symptom score between 8 -35 will be included in this study. Data will be analyzed by SPSS version 23. Descriptive statistics (frequencies, percentages etc.) will be used to describe the socio-demographic characteristics of study population. Independent t-test will be used to compare the mean difference between the groups for AUA score, AMTS score, and pain VAS score. Repeated measure ANOVA will be used to compare the mean score within the group for weekly follow up. Significance level (p value) of the test will be 0.05. Findings of this study will help in establishing incidence of FUS disease and help in estimation of its actual recurrence. This will also help in incorporating IBC in general nursing care for the patients who need it. It will also be helpful in reducing number of OPD visits, length of hospital stay and overall financial burden on health care system.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with diagnosis of urethral stricture.
* Age between 35 - 65 years.
* Females with Body mass index (BMI) < 30.
* Female without any psychiatric illness whose Abbreviated Mental Test Score [AMTS] lies between 7-10.
* Females with moderate to severe urinary symptoms score which lies between 8-35, on American Urological Association (AUA) symptom score.
* Underwent urethral dilation at least once by urologist with subsequent advice of Intermittent Bladder Catheterization (IBC) by trained nurse.
* At presentation >14Fr nelaton catheter could passed per urethra for Intermittent Bladder Catheterization (IBC).
* Female who can read Urdu or English will be included.

Exclusion Criteria:

* Any patient with concomitant bladder or urethral pathology other than urethral stricture.
* Patients unable to perform Intermittent Bladder Catheterization (IBC) due to any physical disability.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 54 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
uretheral stricture recurrence | Total 8 week (every 15 day follow up)
  will be measured by AUA scoring system and visual analogue pain scale

CONTACTS AND LOCATIONS:
Overall Officials: Dr.sabhee UbaidUllah, Study Director — Fauji foundation Lahore cantt
Locations (1):
- UHS, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No